CLINICAL TRIAL: NCT06975306
Title: Radiographic Findings and Clinical Outcomes After Bone Grafting Patellar Defect in ACL Reconstruction
Acronym: BTB BackFill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Anup Shah, Associate Program Director, Orthopaedic Sports Medicine, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005122
Record Dates: First submitted 2025-04-21; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Bone Graft; Complications; ACL Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Grafton demineralized bone matrix gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous bone graft (Experimental): One group will be treated with autologous bone graft for BTB ACLR
  Interventions: Procedure: autologous bone grafts
- Demineralized bone matrix (DBM) putty (Experimental): Demineralized bone matrix (DBM) is a biologic allograft product derived from bone tissue that has undergone a process of demineralization to remove inorganic mineral components while retaining the organic matrix, including proteins and growth factors.
  Interventions: Other: Demineralized bone matrix (DBM)

INTERVENTIONS:
Procedure: autologous bone grafts — group will be treated with autologous bone graft for BTB ACLR
  Arms: autologous bone graft
Other: Demineralized bone matrix (DBM) — Demineralized bone matrix (DBM) is a biologic allograft product derived from bone tissue that has undergone a process of demineralization to remove inorganic mineral components while retaining the organic matrix, including proteins and growth factors.
  Arms: Demineralized bone matrix (DBM) putty

SUMMARY:
All patients will be randomly assigned using a computer randomization algorithm to one of two matched cohort groups. Patients will not be advised which group they belong to until after the completion of the study. One group will be treated with autologous bone graft for bone patellar-tendon bone (BTB) Anterior Cruciate Ligament Reconstruction (ACLR), and the other group will be treated with commercially available DBM (Demineralized bone matrix) putty. Patients will be enrolled from Banner University. Before and after surgery, patient reported outcomes including visual analog pain scale (VAS), Tegner-Lysholm and Cincinnati ACL Test. The principal investigator will evaluate the patients on subjective criteria such as pain and objective criteria including range of motion, arthritic changes seen on radiographs, infection, and ability to kneel.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old,
* male/female/gender neutral,
* all races not including vulnerable/special consideration populations,
* candidate for anterior cruciate ligament reconstruction with bone patellar bone autograft,
* compliant post operative course.

Exclusion Criteria:

* < 18, >41 years of age,
* prior bone patellar bone anterior cruciate ligament reconstruction,
* non-compliance post-operatively,
* nicotine dependence.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
change in surgical time | Duration of Procedure
Change in number of complications from the coring reamer intra-operatively | Duration of Procedure
Change in number of complications associated with displacement of the bone graft | 1 year post procedure
Change in outcomes by immediately filling the patellar void following BTB graft harvest | 1 year post procedure
  Change in outcomes by immediately filling the patellar void following BTB graft harvest, as assessed by the Tegner-Lysholm Knee Scoring Scale
Change in outcomes by immediately filling the patellar void following BTB graft harvest | 1 year post procedure
  Change in outcomes by immediately filling the patellar void following BTB graft harvest, as assessed by the Cincinnati Knee Rating System

CONTACTS AND LOCATIONS:
Overall Officials: Anup Shah, MD, Principal Investigator — College of Medicine - Phoenix
Locations (3):
- United States (3):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Banner Health Center Plus - Arcadia, Phoenix, Arizona
  - Banner Sports Medicine Scottsdale, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schandl K, Horvathy DB, Doros A, Majzik E, Schwarz CM, Csonge L, Abkarovits G, Bucsi L, Lacza Z. Bone-Albumin filling decreases donor site morbidity and enhances bone formation after anterior cruciate ligament reconstruction with bone-patellar tendon-bone autografts. Int Orthop. 2016 Oct;40(10):2097-2104. doi: 10.1007/s00264-016-3246-8. Epub 2016 Jun 29. PMID 27357530
- [Background] Zhang H, Yang L, Yang XG, Wang F, Feng JT, Hua KC, Li Q, Hu YC. Demineralized Bone Matrix Carriers and their Clinical Applications: An Overview. Orthop Surg. 2019 Oct;11(5):725-737. doi: 10.1111/os.12509. Epub 2019 Sep 8. PMID 31496049
- [Background] Leafblad ND, Maak TG. Bone Grafting Technique in Revision ACL Reconstruction: Coring Reamer and Dowel Trick. Arthrosc Tech. 2022 Jun 21;11(7):e1367-e1372. doi: 10.1016/j.eats.2022.03.024. eCollection 2022 Jul. PMID 35936861
- [Background] Tsuda E, Okamura Y, Ishibashi Y, Otsuka H, Toh S. Techniques for reducing anterior knee symptoms after anterior cruciate ligament reconstruction using a bone-patellar tendon-bone autograft. Am J Sports Med. 2001 Jul-Aug;29(4):450-6. doi: 10.1177/03635465010290041201. PMID 11476385
- [Background] Radiological Society of North America (RSNA) and American College of Radiology (ACR). (2022, November 1). Radiation Dose. Radiologyinfo.org. https://www.radiologyinfo.org/en/info/safety-xrayMedical research
- [Background] J. M. Erdal, I. Vik, a. P. Parkar; Bergen/NO & European Society of Radiology. (n.d.). Assessment of effective dose in a series of CT of the knees, time to revise the guidelines? In EPOS. ECR 2016. https://dx.doi.org/10.1594/ecr2016/C-0205
- [Background] Su AW, Hillen TJ, Eutsler EP, Bedi A, Ross JR, Larson CM, Clohisy JC, Nepple JJ. Low-Dose Computed Tomography Reduces Radiation Exposure by 90% Compared With Traditional Computed Tomography Among Patients Undergoing Hip-Preservation Surgery. Arthroscopy. 2019 May;35(5):1385-1392. doi: 10.1016/j.arthro.2018.11.013. Epub 2019 Apr 12. PMID 30987906